CLINICAL TRIAL: NCT02968056
Title: One Staged Hybrid Approach of Minimally Invasively Surgical/Catheter Ablation for Persistent Atrial Fibrillation: A Non-Randomized Controlled Trial
Brief Title: One Staged Hybrid Approach of Surgical/Catheter Ablation for Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ju Mei, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-027
Record Dates: First submitted 2016-11-13; First posted 2016-11-18 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Persistent Atrial Fibrillation
Keywords: atrial fibrillation; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid group (Experimental): Minimally invasive surgical radiofrequency ablation of atrial fibrillation followed by catheterized radiofrequency ablation within the same procedure
  Interventions: Procedure: Radiofrequency ablation
- MIS group (Active Comparator): Minimally invasive surgical radiofrequency ablation of atrial fibrillation only
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency energy is used for ablation in both arms of this study (Hybrid group and MIS group)

SUMMARY:
There are 10 million atrial fibrillation (AF) patients in China, and the patients are risk of stroke, heart failure and sudden death. Persistent AF is still a refractory disease, and single catheter ablation only has a success rate around 30-50%. Hybrid strategy consisting of thoracoscopic epicardial ablation and transvenous endocardial ablation seems to be an attractive procedure to improve the treatment of persistent AF. However, only a few centers reported their preliminary results, and the conclusions are controversial. The investigator previously reported a minimally invasive surgical ablation from left thoracoscope only and achieved good results. Recently, the investigator successfully explored a hybrid procedure combing this unique surgical technique and transvenous catheter ablation. Here, the investigator present a study to evaluate the efficacy and safety of this novel hybrid procedure. The hypothesis is that a hybrid approach is more efficient than surgical ablation alone in the treatment of persistent AF.

This study is a non-randomized controlled study within a single institution. Isolated persistent AF patients admitted to the cardiovascular surgery department of Shanghai Xinhua Hospital will be screened for enrollment of this study. The study will recruit 180 patients in total. Based on their own willingness, the patients will be divided into hybrid group and minimally invasive (MIS) group. The MIS group patients only have surgical ablation surgery from left thoracoscope as the investigator reported before, while the hybrid group patients will have additional transvenous catheter ablation after the surgical ablation is done during the same operation. The ratio of hybrid to MIS group is expected to be 1:1, so that each group contains 90 patients. The perioperative data is collected, and the patients will be followed for 6 months. The primary outcome is the rate of sinus rhythm at 6 months post operation. The secondary outcomes include off antiarrhythmic drug rate, perioperative complications, major cardiovascular events, stroke, left ventricular systolic function, medical expense, serum brain natriuretic peptide level and quality of life. The aim is to evaluate the efficacy and safety of this novel hybrid procedure, therefore to provide more evidence of the hybrid strategy in the treatment of persistent AF.

ELIGIBILITY:
Inclusion Criteria

1. Isolated atrial fibrillation, without structural heart disease.
2. Persistent atrial fibrillation (Af last time > 7 days, including persistent long standing atrial fibrillation)
3. Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication; symptomatic patients are those who have been aware of their AF at any time within the last 5 years before enrolment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of these.
4. Patient admitted with intent to treat by either hybrid or surgical ablation
5. Consent

Exclusion Criteria

1. Previous surgical ablation of atrial fibrillation
2. Concomitant other cardiac diseases which require surgery at the same procedure, such as heart valve disease, congenital heart disease, coronary disease, dilated cardiomyopathy etc.
3. With other forms of severe arrhythmia
4. Ejection fraction of left ventricle less than 30%
5. Anteroposterior diameter of left atrial over 60mm
6. Tumor, active infection, pregnancy.
7. Previous surgeries with left thoracotomy, or expected left pleural adhesion, such as history of tuberculosis infection, pleural effusion, pneumothorax etc.
8. Hyperthyroidism
9. Thrombosis within left atrial appendage
10. General conditions too weak to tolerate the surgeries
11. Patient's circumstance that precludes completion of follow-up and/or obtaining information from the 1-year follow-up
12. Other conditions not appropriate for this study based on the investigators' judgments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Sinus rhythm maintenance rate | At 6 months after the surgery
  Based on ECG results from 3 months and 6 months after the surgery. Any non-sinus rhythm lasting >30 seconds captured on ECG at any time will be considered failure to maintain sinus rhythm

SECONDARY OUTCOMES:
Off any antiarrhythmic drug rate | 6 months after the surgery
  The rate is counted at 6 months
Perioperative complications | Within 1 month after the surgery
  Emergent thoracotomy or exploration for bleeding, renal dysfunction requiring new dialysis treatment, respiratory dysfunction requiring prolonged mechanical ventilation with tracheotomy, new pacemaker implantation, and perioperative death
Major cardiovascular events | Within 6 months after discharge
  Death, Nonfatal myocardial infarction, re-admission because of heart disease
Stroke | Within 6 months after the surgery
  New onset of stroke after the surgery
Left ventricular systolic function | At 6 months after the surgery
  Evaluated by ejection fraction from echocardiogram
Costs of treatment in Chinese Yuan | From surgery to 6 months after the surgery
  There are 3 parts. 1. Cost during the first hospitalization; 2. Cost of all the health care from first discharge to 6 months after the surgery, including seeing clinics, medication, re-hospitalization related to atrial fibrillation/surgical complications/new onset of stroke/other atrial fibrillation related complications. 3. Total cost: the combination of the abovementioned two parts.
Serum brain natriuretic peptide level | 6 months after the surgery
Quality of life | 6 months after the surgery
  Evaluated by short form 36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zhou, MD, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boersma LV, Castella M, van Boven W, Berruezo A, Yilmaz A, Nadal M, Sandoval E, Calvo N, Brugada J, Kelder J, Wijffels M, Mont L. Atrial fibrillation catheter ablation versus surgical ablation treatment (FAST): a 2-center randomized clinical trial. Circulation. 2012 Jan 3;125(1):23-30. doi: 10.1161/CIRCULATIONAHA.111.074047. Epub 2011 Nov 14. PMID 22082673
- [Background] Muneretto C, Bisleri G, Bontempi L, Cheema FH, Curnis A. Successful treatment of lone persistent atrial fibrillation by means of a hybrid thoracoscopic-transcatheter approach. Innovations (Phila). 2012 Jul-Aug;7(4):254-8. doi: 10.1097/IMI.0b013e31826f0462. PMID 23123991
- [Background] Pison L, La Meir M, van Opstal J, Blaauw Y, Maessen J, Crijns HJ. Hybrid thoracoscopic surgical and transvenous catheter ablation of atrial fibrillation. J Am Coll Cardiol. 2012 Jul 3;60(1):54-61. doi: 10.1016/j.jacc.2011.12.055. PMID 22742400
- [Background] Pokushalov E, Romanov A, Elesin D, Bogachev-Prokophiev A, Losik D, Bairamova S, Karaskov A, Steinberg JS. Catheter versus surgical ablation of atrial fibrillation after a failed initial pulmonary vein isolation procedure: a randomized controlled trial. J Cardiovasc Electrophysiol. 2013 Dec;24(12):1338-43. doi: 10.1111/jce.12245. Epub 2013 Sep 9. PMID 24016147
- [Background] Cox JL. A brief overview of surgery for atrial fibrillation. Ann Cardiothorac Surg. 2014 Jan;3(1):80-8. doi: 10.3978/j.issn.2225-319X.2014.01.05. PMID 24516803
- [Background] Gelsomino S, Van Breugel HN, Pison L, Parise O, Crijns HJ, Wellens F, Maessen JG, La Meir M. Hybrid thoracoscopic and transvenous catheter ablation of atrial fibrillation. Eur J Cardiothorac Surg. 2014 Mar;45(3):401-7. doi: 10.1093/ejcts/ezt385. Epub 2013 Jul 31. PMID 23904136
- [Background] Mei J, Ma N, Ding F, Chen Y, Jiang Z, Hu F, Xiao H. Complete thoracoscopic ablation of the left atrium via the left chest for treatment of lone atrial fibrillation. J Thorac Cardiovasc Surg. 2014 Jan;147(1):242-6. doi: 10.1016/j.jtcvs.2012.10.005. Epub 2012 Nov 2. PMID 23122696
- [Background] Pragliola C, Mastroroberto P, Gaudino M, Chello M, Covino E. Staged transthoracic approach to persistent atrial fibrillation (TOP-AF): study protocol for a randomized trial. Trials. 2014 May 26;15:190. doi: 10.1186/1745-6215-15-190. PMID 24885377
- [Background] Bulava A, Mokracek A, Hanis J, Kurfirst V, Eisenberger M, Pesl L. Sequential hybrid procedure for persistent atrial fibrillation. J Am Heart Assoc. 2015 Mar 25;4(3):e001754. doi: 10.1161/JAHA.114.001754. PMID 25809548
- [Background] Wang PJ. Hybrid epicardial and endocardial ablation of atrial fibrillation: is ablation on two sides of the atrial wall better than one? J Am Heart Assoc. 2015 Mar 25;4(3):e001893. doi: 10.1161/JAHA.115.001893. No abstract available. PMID 25809549
- [Background] Beukema RJ, Adiyaman A, Smit JJ, Delnoy PP, Ramdat Misier AR, Elvan A. Catheter ablation of symptomatic postoperative atrial arrhythmias after epicardial surgical disconnection of the pulmonary veins and left atrial appendage ligation in patients with atrial fibrillation. Eur J Cardiothorac Surg. 2016 Jan;49(1):265-71. doi: 10.1093/ejcts/ezv047. Epub 2015 Feb 26. PMID 25721819
- [Background] Phan K, Phan S, Thiagalingam A, Medi C, Yan TD. Thoracoscopic surgical ablation versus catheter ablation for atrial fibrillation. Eur J Cardiothorac Surg. 2016 Apr;49(4):1044-51. doi: 10.1093/ejcts/ezv180. Epub 2015 May 23. PMID 26003961
- [Background] Richardson TD, Shoemaker MB, Whalen SP, Hoff SJ, Ellis CR. Staged versus Simultaneous Thoracoscopic Hybrid Ablation for Persistent Atrial Fibrillation Does Not Affect Time to Recurrence of Atrial Arrhythmia. J Cardiovasc Electrophysiol. 2016 Apr;27(4):428-34. doi: 10.1111/jce.12906. Epub 2016 Jan 29. PMID 26725742
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422